CLINICAL TRIAL: NCT06593509
Title: The Effectiveness of High Flow Nasal Cannula Versus Noninvasive Ventilation and Conventional Oxygen Therapy in Patients Weaned from Invasive Mechanical Ventilation:
Brief Title: The Effectiveness of High Flow Nasal Cannula Versus Noninvasive Ventilation and Conventional Oxygen Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 443/2023
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Post Extubation Respiratory Failure
Keywords: weaning.; Mechanical ventilation; COT; HFNC; NIV

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Non-invasive mechanical ventilation (Experimental): Device: Non-invasive mechanical ventilation Bilevel pressure support through a face mask
  Interventions: Device: Maquet,Servo I.
- High Flow Conditioned Oxygen Therapy (Experimental): Device: High Flow Conditioned Oxygen device vapotherm via nasal cannula
  Interventions: Device: Vapotherm
- Conventional Oxygen Therapy (Active Comparator): Device: Conventional Oxygen Therapy conventional Oxygen Therapy with Venturi facial mask.
  Interventions: Device: venturi mask

INTERVENTIONS:
Device: Maquet,Servo I. — Model number: 06487800, Serial Number: 19761, SKU#: Inv-00344191, Made in Sweden
  Arms: Non-invasive mechanical ventilation
Device: Vapotherm — INC ,100 domain drive Exeter, NH 03833, Made in U.S.A
  Arms: High Flow Conditioned Oxygen Therapy
Device: venturi mask — Intersurgical Ltd, Crane House, Molly Millars Lane, Wokingham, Berkshire, RG41 2RZ, UK.,REF. 1107085, LOT,31757961
  Arms: Conventional Oxygen Therapy

SUMMARY:
A prospective, randomized controlled study enrolling sixty patients who fulfilled weaning criteria after requiring invasive MV. After extubation, patients were randomized into three groups (20 patients per group) :NIV group , HFNC group, and COT group. Primary outcomes included reintubation rates at certain time points and after 48 hours post-extubation while secondary outcomes included time to reintubation , ICU length of stay, ICU mortality. Objective: To compare the rate of reintubation within 48 hours after extubation among patients receiving NIV, HFNC and COT as post-extubation respiratory support.

DETAILED DESCRIPTION:
Reintubation after liberation from mechanical ventilation (MV) is a wellknown adverse event seen in different patients subtypes(post surgical, trauma,medical) as well as in surgical and medical intensive care units (ICUs) .The cumulative probability of reintubation , following planned and unplanned extubation , in 185 ICUs in the United States ,reached up to 10 % and 90% occurred within the first 96 hours (4 days) after first extubation , the median time to reintubation was 15 hours.

Proper timing for extubation is crucial to minimize extubation failure and about 12 to 14% of patients planned for extubation would require reintubation within 48 to 72 hours, mostly within the first 24 hours & in a multivariate analysis, duration of MV more than 7 days prior to extubation, ineffective cough, and severe systolic left ventricular dysfunction were independent factors associated with extubation failure, whereas ,in another study,age and underlying diseases were other factors associated with higher extubation failure with rates reaching up to 34% in patients 65 yrs or older, those with chronic respiratory or cardiac disorders and the condition was specifically associated with significant rapid clinical deterioration and worsening of daily organ dysfunction scores reflecting a direct effect of reintubation on patient outcomes. Mortality risk is reported to be five times higher in patients who require reintubation after extubation from MV.

Postextubation sequential oxygen devices applied as first-line therapy after extubation include noninvasive ventilation (NIV) , high-flow nasal cannula (HFNC) and conventional oxygen therapy (COT).

COT delivered via masks and nasal prongs has been widely used as the main sequential supportive oxygen therapy administered to patients after extubation . However, the maximal oxygen flow rates that these devices can deliver are limited with maximum flow rate up to 15 L/min only, which is usually far lower than the demands that postextubation patients would require . The fraction of inspired oxygen (FiO2) delivered by COT is unstable because of the entertainment of room air and dilution of the inspired oxygen .

Potential benefits of NIV include the ability to provide a relatively consistent and wider range of FiO2 compared with COT . Moreover, NIV creates an extrinsic positive end expiratory pressure which aids in recruitment of collapsed alveoli.

The American College of Chest Physicians/American Thoracic Society (ACCP/ATS) clinical practice guidelines for liberation from MV in the critically ill highlight the importance of usage of preventive (NIV) in patients at high risk of reintubation and emphasizing its impact on improving oxygenation, ventilation, decreasing hospital mortality, length of hospital stay, and incidence of ventilator associated pneumonia (VAP) . Evidence suggest that NIV may prevent postextubation respiratory failure and avoid reintubation if it is applied soon after extubation. On the other hand, this strategy is associated with worse outcomes if applied after development of postextubation acute respiratory failure (ARF). In addition, intolerance to NIV is quite common in clinical practice, eye irritation, skin damage, interruption in diet and clearance of airways secretion are common adverse events and can worsen the patient's outcome. These limitations urge investigators to explore other alternative oxygen delivery devices and search for potential roles in improving clinical outcomes in the post extubation setting.

High flow nasal cannula (HFNC) is a novel, high flow oxygen device with established efficiency, it is well tolerated by patients, easily applied and can provide fully humidified, heated, high-flow rates up to 60 L/min, a constant high fraction of inspired oxygen (FiO2) (0.21 - 1.0) and flow-dependent continuous positive airway pressure (2-5 cm H2O) which , in turn , increases end-expiratory lung volume and aids in alveolar recruitment and reduces atelectasis, subsequently improving ventilation-perfusion mismatch . The continuous high flow of oxygen guarantees both higher tidal volume with adequate minute ventilation and sufficient oxygenation improves inspiratory flow dynamics and decrease work of breathing by improving thoracoabdominal synchrony. In addition, pharyngeal dead space washout effect decreases carbon dioxide in a faster manner. Finally, the heated humidification flow creates physiological conditions preserving mucosal integrity, reducing mucosal inflammation, and facilitating clearance of secretions, thereby improving the oxygenation, and further decreasing the risk of atelectasis.

Several studies have investigated these available devices and compared their efficacy in lowering reintubation rates after extubation, but results are conflicting and inconsistent and no study could conclude that either HFNC, NIV or COT is superior to prevent reintubation. One randomized controlled trial (RCT) reported that HFNC was associated with a lower rate of reintubation in low-risk patients compared to COT. Another RCT in high-risk non-hypercapnic patients and concluded that HFNC could not decrease rate of reintubation compared with COT. A third study showed that HFNC and NIV are equally effective in lowering reintubation rate.

In Egypt, researchers have also studied and compared the effectiveness of these modalities in different clinical ICU settings with comparable efficacies between three devices. The objective of the current work is to compare the rate of reintubation after extubation using HFNC versus NIV and COT as sequential respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years)
* who were mechanically ventilated longer than 12 hours for various respiratory indications
* and planned for liberation from MV after fulfilling the criteria for weaning

Exclusion Criteria:

* patients (<18 years )
* Tracheostomized patients,
* patients who were self-extubated or accidentally extubated,
* Presence of contraindication to NIV : facial trauma, fracture or burn, pneumothorax, bronchopleural fistula, gastro/esophageal bleeding,
* and patients who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
reintubation rate(N,%) | 48 hours
  reintubation after extubation

SECONDARY OUTCOMES:
intensive care unit length of stay(days) | one month
  duration of stay in intensive care unit
intensive care unit mortality rate(N,%) | one month
  mortality inside intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Emad Eldine A korraa, MD, Study Director — chest department ,ain shams university,cairo,egypt; Rehab M Mohammad, MD, Principal Investigator — chest department ,ain shams university,cairo,egypt; amira AA elghonemy, M.B.B.Ch, Principal Investigator — chest department ,ain shams university,cairo,egypt
Locations (1):
- Respiratory intensive care unit , chest department faculty of medicine ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No